CLINICAL TRIAL: NCT01404273
Title: Functional MRI of an Open Trial of Relaxation Response Training in Adults With Attention-Deficit/Hyperactivity Disorder
Brief Title: Functional MRI of Relaxation Response Training in Adults With Attention-Deficit/Hyperactivity Disorder
Acronym: ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, George Bush, Director of Neuroimaging Research, Benson-Henry Institute for Mind-Body Medicine at MGH, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009P002052
Record Dates: First submitted 2011-07-25; First posted 2011-07-28 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Meditation

ARMS (1):
- Meditation/Relaxation Response Training (Experimental)
  Interventions: Behavioral: Meditation/Relaxation Response Training

INTERVENTIONS:
Behavioral: Meditation/Relaxation Response Training — 1 hour weekly sessions with 20 min daily home practice for 6 weeks

SUMMARY:
This research study is being done to examine how meditation and the relaxation response (RR) may change brain activity in attention-deficit/hyperactivity disorder (ADHD).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults (ages 18 - 49).
2. Patients with the diagnosis of Attention Deficit Hyperactivity Disorder (ADHD), by the Diagnostic and Statistics Manual of Mental Disorders (DSM-IV), as manifested in clinical evaluation and confirmed by structured interview.

Exclusion Criteria:

1. Any current, non-ADHD Axis I psychiatric conditions
2. Baseline Beck Depression Inventory (BDI) > 19.
3. Any clinically significant chronic medical condition.
4. Mental retardation
5. Organic brain disorders
6. Seizures or tics.
7. Pregnant or nursing females.
8. Clinically unstable psychiatric conditions (suicidal behaviors, psychosis).
9. Current or recent (within the past 2 years) substance abuse or dependence.
10. Patients currently or recently (within past 1 month) on psychotropic medication.
11. Subjects with current or prior adequate psychopharmacologic treatment for ADHD.
12. Regular practice of an Relaxation Response-inducing technique within the past year
13. History of claustrophobia or any of the standard contraindications to magnetic resonance imaging (MRI) scanning(metal objects within body).

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change in functional magnetic resonance imaging (fMRI) activation from baseline after a 6-week intervention | 2 sessions, 2 hours each to be conducted before and after the 6-week intervention
  functional magnetic resonance imaging (fMRI) activation in dorsal anterior medial cingulate cortex (daMCC) & dorsolateral prefrontal cortex (DLPFC) during multi-source interference task (MSIT)

CONTACTS AND LOCATIONS:
Overall Officials: George Bush, M.D., Principal Investigator — MGH
Locations (1):
- Benson-Henry Institute, 151 Merrimac St, 4th Floor, Boston, Massachusetts, United States